CLINICAL TRIAL: NCT04316910
Title: Characterisation of Gut Microbiota in Patients Undergoing Gastrointestinal Surgery With Postoperative Delirium (GIM-POD)
Acronym: GIM-POD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Wen-fei Tan, clinical professor, China Medical University, China
Other Study IDs: 20200319
Record Dates: First submitted 2020-03-19; First posted 2020-03-20 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Delirium; Gut Microbiota
MeSH Terms: conditions — Emergence Delirium | interventions — Anesthetics, General

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative delirium: The CAM-ICU (Confusion Assessment Method for Intensive Care Unit) was used for delirium assessment.
  Interventions: Drug: General anesthetic
- Non-Postoperative delirium: The CAM-ICU (Confusion Assessment Method for Intensive Care Unit) was used for delirium assessment.
  Interventions: Drug: General anesthetic

INTERVENTIONS:
Drug: General anesthetic — General anesthesia was induced as follows: 0.3 mg kg-1 intravenous (IV) etomidate, 2 mg IV midazolam, 0.4 μg kg-1 IV sufentanil, and 0.2 mg kg-1 IV cisatracurium. Anesthesia was maintained with an end-tidal concentration of 2-3 vol% sevoflurane and 0.2-0.3 μg kg-1h-1 sufentanil to maintain the bispectral index between 40 and 60.

SUMMARY:
The study is a case-controlled observational trial. Sixty patients will be divided into 2 groups depending on whether postoperative delirium or not. This study aims to characterise the gut microbiota in patients undergoing gastrointestinal surgery with postoperative delirium. The CAM-ICU (Confusion Assessment Method for Intensive Care Unit) was used for delirium assessment.

DETAILED DESCRIPTION:
The study is a case-controlled observational trial. Sixty patients will be divided into 2 groups depending on whether postoperative delirium or not. This study aims to characterise the gut microbiota in patients undergoing gastrointestinal surgery with postoperative delirium. The CAM-ICU (Confusion Assessment Method for Intensive Care Unit) was used for delirium assessment.

General anesthesia was induced as follows: 0.3 mg kg-1 intravenous (IV) etomidate, 2 mg IV midazolam, 0.4 μg kg-1 IV sufentanil, and 0.2 mg kg-1 IV cisatracurium. Anesthesia was maintained with an end-tidal concentration of 2-3 vol% sevoflurane and 0.2-0.3 μg kg-1h-1 sufentanil to maintain the bispectral index between 40 and 60.

ELIGIBILITY:
Inclusion Criteria:

* 1. ethnic Chinese;
* 2. age, 18 to 80 years old;
* 3. American Society of Anaesthesiologists (ASA) physical status I or II;
* 4. required Gastrointestinal Surgery

Exclusion Criteria:

* Cognitive difficulties
* Partial or complete gastrectomy
* Previous esophageal surgery
* Previous treated by radiotherapy or surgery
* Inability to conform to the study's requirements
* Deprivation of a right to decide by an administrative or juridical entity
* Ongoing participation or participation in another study <1 month ago

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients Undergoing Gastrointestinal Surgery
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-07-19 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Characterisation of Gut Microbiota | from baseline to postoperative 72 hours
  this study will characterise gut microbiota in 2 groups of 30 patients

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of China Medical University, Shenyang, Liaoning, China